CLINICAL TRIAL: NCT04215432
Title: Effect of Propolis Extract, Nanovitamin C and Nanovitamin E in Clinical and Microbiological Parameters of Peri-implant Mucositis: A Double-blind, Randomized, Clinical Trial
Brief Title: Propolis Extract, Nanovitamin C and Nanovitamin E in Peri-implant Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Bio Nature Essences S.L (Unknown)
Responsible Party: Principal Investigator, Rosa María López-Pintor Muñoz, Associate professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0004
Record Dates: First submitted 2019-12-21; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Peri-implant Mucositis
Keywords: dental implants; peri-implant mucosits; toothpaste; propolis; nanovitamin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Test group (Experimental): Gel contained in tubes with the same appearance (30g), identical in colour, flavour and density, with the following components: Sodium-Monofluorophosphate, Silicon Dioxide, Glycerin, D-sorbitol, Polyethylene glycol, Sodium Carboxymethylcellulose, Xylitol, Sterol Glycoside, Peppermint Oil, L-Menthol, Methyl Hydroxybenzoate, Deionized Water, Propolis Extract (2%), Ascorbic Acid (0.2%) and Tocopherol Acetate (0.2%).
  Interventions: Device: Gel containing propolis extract, nanovitamin C and nanovitamin E
- Placebo group (Placebo Comparator): Gel contained in tubes with the same appearance (30g), identical in colour, flavour and density, with the following components: Sodium-Monofluorophosphate, Silicon Dioxide, Glycerin, D-sorbitol, Polyethylene glycol, Sodium Carboxymethylcellulose, Xylitol, Sterol Glycoside, Peppermint Oil, L-Menthol, Methyl Hydroxybenzoate, Deionized Water and E155/151 coloring.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Gel containing propolis extract, nanovitamin C and nanovitamin E — The patient had to use the gel as a toothpaste and apply it with an interdental brush in mesial and distal aspects of the implant with peri-implant mucositis. during 1 month.
  Arms: Test group
Device: Placebo — The patient had to use the gel as a toothpaste and apply it with an interdental brush in mesial and distal aspects of the implant with peri-implant mucositis.
  Arms: Placebo group

SUMMARY:
The objective of this study was to perform the first clinical trial to evaluate the effectiveness of propolis extract, nanovitamin C and nanovitamin E gel as adjuvant to mechanical debridement in clinical and microbiological parameters of implants with peri-implant mucositis

ELIGIBILITY:
Inclusion Criteria:

* cooperative adult patients,
* with one or more implants with peri-implant mucositis, and
* presenting at least 18 months of functional loading.

Exclusion Criteria:

* refuse to participate in the study,
* patients who had implants with peri-implantitis (BOP and/or suppuration together with progressive radiographic marginal bone loss),
* patients with uncontrolled periodontitis (presence of nine or more sites with PD ≥ 5 mm and with full-mouth bleeding score (FMBS) > 25%),
* systemic diseases or conditions that could alter the results of the study (diabetes mellitus, immunosuppression, infectious diseases, rheumatoid disease, history of bisphosphonate treatment, radiotherapy, chemotherapy, etc.),
* patients who had taken local and/or systemic antibiotics less than 2 months ago,
* pregnant or breastfeeding women, and
* patients with history of allergies to the test and/or placebo components administered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Changes in bleeding on probing | baseline and 1-month follow-up
  It was present when it appeared bleeding at the gingival margin after recording probing depths at six sites in each implant. Modified bleeding index was also collected.

SECONDARY OUTCOMES:
Changes in probing depth | baseline and 1-month follow-up
  It was recorded at six sites of each implant with PM, using a probe with a force of 0.2N (PCV12; HuFriedy, Chicago, IL, EEUU).
Changes in plaque index | baseline and 1-month follow-up
  It was recorded after using a disclosing dye, as the presence of dental plaque at the gingival margin at six sites in each implant.
Changes in microbilogical sample | baseline and 1-month follow-up
  Microbiological samples were obtained at the deepest peri-implant pocket. Firstly, the area was isolated using cotton rolls and dried with a gentle air blow. Then, three sterile paper tips (#30, Maillefer, Ballaigues, Switzerland) were left for 10 seconds at the point with the greatest peri-implant pocket depth. Finally, the papers were introduced in a vial containing 1.5 ml of reduced transport fluid.
  The vials were sent to the microbiology laboratory of the School of Dentistry, at Complutense University of Madrid for an anaerobic culture within 24 hours. Total counts and counts of target periodontal pathongens [Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Prevotella intermedia, Tannerella forsythia, Parvimonas micra, Fusobacterium nucleatum, Campylobacter rectus, Eikenella corrodens, Capnocytophaga sp., Actinomyces odontolyticus] were determined after 7-14 days of anaerobic incubation. Then, those results were converted in colony-forming units per ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided